CLINICAL TRIAL: NCT02253498
Title: The Safety and Efficacy of Long-term Treatment of PINS Stimulator System for Tourette Syndrome
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Pins Medical Co., Ltd (Industry)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PINS-009
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-05

CONDITIONS: Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Deep Brain Stimulation (Experimental): Deep Brain Stimulation is on
  Interventions: Device: deep brain stimulation (DBS)
- Sham Stimulation (Sham Comparator): placebo
  Interventions: Device: deep brain stimulation (DBS)

INTERVENTIONS:
Device: deep brain stimulation (DBS)
  Other Names: Implanted device

SUMMARY:
The purpose of this clinical study is to verify the long term effectiveness and safety of a bilateral deep brain stimulation (DBS) produced by Beijing PINS Medical Co., Ltd. as a treatment option for patients with cognitive, behavioral, and functional disability of Tourette Syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is aged 18 or older
2. Patient Group with Tourette's syndrome, Diagnosis of Tourette Syndrome by DSM-IV

Exclusion Criteria:

1. Major Depressive Episode within the previous 6 months
2. Schizophrenia or other psychotic disorder.Participate in other clinical trial;
3. Has a life expectancy of < 1 year.
4. The investigator and/or enrollment review committee, would preclude participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Modified Rush Video Rating Scale (mRVRS) | 12 month

SECONDARY OUTCOMES:
Tourette Syndrome Symptom List (TSSL) | 12 month
SF-36 | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Li Luming, PhD, Study Chair — Tsinghua University